CLINICAL TRIAL: NCT01698710
Title: EUS Guided Injection of Albumin Bound Paclitaxel Into Pancreatic Cysts
Brief Title: Endoscopic Abraxane Injection Into Pancreatic Cysts
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: expiration of IRB approval
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, William R. Brugge, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-178
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2014-09

CONDITIONS: Pancreatic Cysts
Keywords: Premalignant; Malignant
MeSH Terms: conditions — Pancreatic Cyst; Precancerous Conditions | interventions — Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Albumin bound paclitaxel (Experimental): Albumin bound paclitaxel will be administered into the mucinous cyst of pancreas in endoscopy procedure.
  Interventions: Drug: Albumin bound paclitaxel

INTERVENTIONS:
Drug: Albumin bound paclitaxel — Albumin bound paclitaxel will be administered into the mucinous cyst of pancreas in endoscopy procedure.
  Other Names: Abraxane

SUMMARY:
This research study is a pilot study. In this pilot study we are testing the safety of a procedure. "Investigational" means that the Albumin bound paclitaxel (Abraxane) is still being studied and that research doctors are trying to find out more about it. It also means that the FDA has not approved Abraxane injection for your type of medical condition. Treatment of pancreatic cysts often requires follow-up imaging studies and surgical resection of the cysts. As part of standard medical care, you will be undergoing a diagnostic endoscopic ultrasound guided fine needle aspiration (EUS-FNA) in order to evaluate type of the cyst. During the EUS and just after the cyst fluid aspiration, you will undergo the injection of the drug into the cyst cavity if your cyst is thought to be cancerous or precancerous. Cyst fluid will be analyzed for further diagnosis.

DETAILED DESCRIPTION:
You will be asked to undergo some screening tests or procedures to find out if you can be in the research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated. Screening tests include the following: medical history, performance status, assessment of pancreatic cyst by CT, MRI or EUS, blood tests and a pregnancy test.

If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria you will not be able to participate in this research study.

As part of your medical care you will be undergoing an endoscopic procedure EUS-FNA (Endoscopic Ultrasound Fine Needle Aspiration) in order to evaluate and evacuate the cyst fluid. During the EUS-FNA and just after the cyst fluid aspiration, albumin bound paclitaxel will be injected into the cyst cavity.

The study procedure (injection of drug into cyst cavity) takes place over 5 minutes during the EUS-FNA. 2 days after the procedure you will receive a phone call from the research coordinator to check on how you are feeling. 3 months after study procedure participants will undergo a follow up CT to see what happened to the cyst. You will continue to have routine follow up for your medical problems.

ELIGIBILITY:
Inclusion Criteria:

* Mucinous cysts (premalignant or malignant cysts of the pancreas)
* Normal organ and marrow function
* Baseline CT within 6 months of enrollment

Exclusion Criteria:

* Pregnant or breastfeeding
* Acute active pancreatitis
* Complicated pancreatic cysts
* Subjects who do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Brugge, MD, Principal Investigator — Massachusetts General Hospital

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Albumin Bound Paclitaxel
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Albumin Bound Paclitaxel
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5
Cyst diameter [Mean (Full Range); unit: mm] — Patients with clinically diagnosed mucinous cysts (premalignant or malignant cysts of the pancreas) including mucinous cystic neoplasms and intraductal papillary mucinous neoplasms were eligible.
  mm | 28.4 [23 to 35]
Location of cyst [Count of Participants; unit: Participants] — Patients with clinically diagnosed mucinous cysts (premalignant or malignant cysts of the pancreas) including mucinous cystic neoplasms and intraductal papillary mucinous neoplasms were eligible.
  Participants
    Head | 4
    Body | 1

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Pancreatitis
Description: Safety of injection of albumin-bound paclitaxel will be measured by the frequency of pancreatitis.
Time Frame: 3-10 months (median 6 months) after injection therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin Bound Paclitaxel
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Feasibility of Endoscopic Ultrasonography (EUS) Guided Injection of Albumin-bound Paclitaxel Into Pancreatic Cysts
Description: The feasibility of the procedure will be measured by the ease of injection of albumin-bound paclitaxel into the cyst cavity across the gastro-duodenal wall. On a subjective scale, the endoscopist will note the ease of the procedure on a scale of 0-5, with 5 being very easy and 0 is not possible. Any score less than 2 will be considered unacceptable and failure of the study.
Time Frame: immediately after procedure
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Albumin Bound Paclitaxel
Number analyzed (Participants) | 5
units on a scale | 4 [3 to 5]

3. Secondary Outcome: Size of Cystic Lesion
Description: Determine the size of the cystic lesion using CT scanning. Number of participants with reduction in size, persistent size, or increase in size of cyst are reported.
Time Frame: 3-10 months (median 6 months) after injection therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Albumin Bound Paclitaxel
Number analyzed (Participants) | 5
Participants
  Reduction | 3
  Persistent | 1
  Increase | 1

ADVERSE EVENTS:
Arm/Group | Albumin Bound Paclitaxel
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes